CLINICAL TRIAL: NCT03933540
Title: Evaluating the Association Between Activity and PROMIS Pediatric Measures in Children With Chronic Conditions
Brief Title: Association Between Activity and PROMIS Pediatric Measures in Children With Asthma
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00100297
Record Dates: First submitted 2019-04-26; First posted 2019-05-01 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-02

CONDITIONS: Pediatric Asthma
Keywords: Patient Reported Outcome Measures; Activity Monitors; Pedometry; PROMIS; Health Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Asthma Patients: Participants are ages 8 years through 17 years and have partially controlled or uncontrolled asthma.
  No intervention is included in this study.

SUMMARY:
Aim: Determine the association between activity (steps taken) and PROMIS Pediatric measures in order to explore the use of pedometry data to augment PROs in research and clinical care.

The investigators will evaluate the associations between activity trackers and scores on PROMIS pediatric measures in adolescents with partially controlled or uncontrolled asthma, aged 8 through 17 years. The investigators hypothesize that daily step data will be highly correlated with and responsive when measured against PROMIS Pediatric measures of Physical Activity and Physical Function-Mobility.

The Asthma (not well controlled) cohort will receive Garmin Vivofit3 activity monitors in clinic/and or home and wear them continuously for 4 weeks while completing PROMIS measures, the ecological survey, and an additional asthma control survey online (from home) via the PRO-Core data collection system at the end of each of those 4 weeks. They will return the Vivofit3 in a follow up clinic/and or home visit at the end of the 4 week period. In addition, children/adolescents will complete a spirometry test at baseline and follow up clinic/home visits. Written and verbal instructions for Vivofit3 use will be provided. Trained CRAs will communicate frequently with participants, including when the monitor is received by the participant and when the monitors need to be returned. Monitor data will be uploaded to the device user account in the Garmin Connect Mobile App by the CRA upon return of the monitor. Data from device user accounts will be imported into a UNC PRO-Core study database. Asthma participants will receive $20 at each of the two clinic/and or home visits and $10 per completed survey.

Measures and Analyses: Cross-sectional analyses of daily step and PROMIS Pediatric measures will be used to test convergent validity of conceptually linked measures. Results from regression models for longitudinal data analyses of PRO measures will be benchmarked against regression results from step data, to ascertain responsiveness. The investigators will use descriptive statistics to understand patterns by condition; the investigators will analyze data in aggregate and test whether disease group (covariate) is associated with outcomes. Analyses will control for demographics, mental health, and ecologic factors such as sports participation and season/weather.

Risk/Safety issues: This is a minimal risk study. Participants may be at risk for skin irritation due to continual monitor wear. Additionally, there is always a risk of breach of confidentiality associated with all research.

DETAILED DESCRIPTION:
Purpose of the study:

The investigators will evaluate the associations between activity trackers and scores on PROMIS pediatric measures in adolescents with partially controlled or uncontrolled asthma, aged 8 through 17 years. The investigators hypothesize that daily step data will be highly correlated with and responsive when measured against PROMIS Pediatric measures of Physical Activity and Physical Function-Mobility.

The knowledge gained in this study could have direct clinical benefits, such as it will allow us to determine the association between steps taken (pedometer data) and PROMIS Pediatric measures in order to explore the use of pedometry data to augment PROs in future research and clinical care or to serve as a proxy measure for patients who are not able to self-report due to limitations in language, literacy, cognition or health status. Based on prior work with other PRO measures 18-20, the investigators expect that increased daily and weekly step numbers will reflect better overall health status. Pedometry may prove to be a useful proxy for health status in future research studies when adolescents are too ill to self-report using PROMIS or other traditional PROs.

Background and Significance:

Patient Reported Outcome (PRO) measures provide the opportunity to more fully gauge response to disease and therapy, providing actionable health information to take treatment to a more personalized level. For PRO measures to be widely adopted for use in either clinical trials 1 or by health care providers, there must be substantial evidence for the reliability and validity of the PRO measure in the specific population. One of the most essential aspects of the appropriateness of a PRO measure is documentation of the responsiveness of the PRO measure, which indicates the ability of the PRO measure to detect change over time when it is expected.

The PROMIS® measures represent a robust set of questionnaires for capturing the patient's experience and have undergone extensive psychometric evaluation. However, PRO measures are subjective and depend on a variety of patient level variables, including the patient's cognition, literacy, language, or health status. Additionally, some situations exist in which children or their parents may not be able to self-report symptoms using PROs due to language barriers, literacy level, or disease activity (too fatigued, etc.). Objectively reported steps, collected via pedometer wear, may be a way to augment the data that the investigators get from PRO measures and to bypass some patient level variables that can affect PRO data.

Pedometers have been shown to be suitable for assessing step activity in children age 6 years and up. A 7-day monitoring period using pedometers provided an accurate estimate of normal physical activity in children and adolescents. Prior research in children has shown correlations between physical activity and psychosocial indicators,4 physical health,5 and cognitive function6; however, there is a deficiency of knowledge related to physical activity in children with chronic illnesses, such as cancer, rheumatic disease, and asthma, association with daily steps, and impacts on health outcomes.

A review of several small pilot studies of physical activity monitoring in adult patients with cancer found physical activity, particularly the number of daily "steps", varied considerably across phases of disease and treatment type, including healthy controls, surgical resection with curative intent, and palliative chemotherapy and palliative radiation.7 Low fitness and decreased exercise capacity have been demonstrated in children with cancer,8 JIA9, 10 and SLE.11 Children with moderate to severe asthma have been shown to get less physical activity than their healthy peers.14, 15 More specifically, children with asthma tend to participate in less moderate to high intensity activity16 and to take fewer daily steps16, though there appears to be little difference in sedentary time for children with asthma and healthy controls.15, 16 However, uncertainties remain regarding the relationships between daily activity levels, disease activity, and relevant domains including physical function, pain interference, fatigue, anxiety and depression.

Design & procedures:

This is a single arm, observational study of 100 patients with partly controlled or uncontrolled asthma. The primary purpose of this study is to determine the association between activity (steps taken) and PROMIS Pediatric measures in order to explore the use of pedometry data to augment PROs in research and clinical care. The investigators anticipate 12 months of participant accruals.

Subjects will participate in two clinic/and or home visits and complete electronic surveys from home at three time points. During the clinic/home visits on Day 0 and Day 28 (+/- 2 days), participants will complete the GINA checklist, a medication review, a spirometry test, have BMI obtained, and complete the Child Asthma Control Test (if 11 years old or younger) or the Asthma Control Test (if 12 years or older). On Day 0, parents will also complete a demographics form and the child participant will recieve their Vivofit3 monitor. The Vivofit3 will be worn 24 hours a day for 4 weeks. At Day 28, CRA's will sync the data from the Vivofit3 monitor to the participants study specific user account in the Garmin Connect Mobile app.

In between Days 0 and 28 participants will complete three sets of electronic surveys. Participants will complete their first set of surveys after 7 full days of VivoFit3 wear (study Day 7), and every 7 days after that (Study days 14, 21, and 28) by clicking on a link in the survey email that will take them to the PRO-Core data collection system. They may complete these surveys from home or anywhere they would like where they have internet access. The Day 28 survey will be completed in clinic/and or home.

The Subject Population:

The study sample (N=100) comprises 50 children between the ages of 8 and 12 and 50 children between the ages of 13 and 17 who have uncontrolled or partly-controlled asthma. The University of North Carolina (UNC) will accrue 30 children in each age group and the Boston site will accrue 20 participants in each age group. Duke is the data coordinating center for this study and will not be recruiting patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 8 to < 18 years
* Patient meets one of the following criteria at the time of screening:

  1. FEV1 (Forced expiratory volume) less than 80% predicted, or
  2. One or more exacerbations requiring systemic steroids in the last year, or
  3. Partly controlled or uncontrolled asthma, using the GINA 2016 guidelines for asthma diagnosis and management
* Ability to read and understand English.
* Provide informed written assent and receive informed written consent from parent.
* Ability and willingness to participate in all study activities, including completion of online surveys and wearing an activity monitor on the wrist for four weeks.
* Ability and willingness to participate in a follow up visit in the clinic/and or home 26 - 30 days after the initial clinic/and or home visit.
* Access to a smart phone, computer, tablet, or other device with internet access that is capable of supporting survey completion via the PRO-Core website.

Exclusion Criteria:

* Clinically significant cognitive or memory impairment in the opinion of clinical or research staff
* A child or adolescent who is under the legal custody of a state or a subdivision of the state.
* Comorbid conditions that could confound results such as chronic heart disease, cystic fibrosis, VCD, etc., as determined by site investigator

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study sample (N=100) comprises 50 children between the ages of 8 and 12 and 50 children between the ages of 13 and 17 who have uncontrolled or partly-controlled asthma.
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Average daily steps | 1 week average, derived for each of the 4 weeks a participant wears the activity monitor for the month of study enrollment.
  Average number of steps per day within a 1 week period, derived from Garmin VivoFit 3 activity monitor data

SECONDARY OUTCOMES:
Self-Reported Asthma Symptoms | Weekly assessment taken at the end of each of the four study weeks.
  Patients rate their asthma symptom severity on a 6 point likert scale ranging from very bad to very good.
PROMIS Pediatric Short Form v2.0 - Asthma Impact | 7 day recall period, taken at the end of each of the four study weeks
  Short form questionnaire assessing impact of asthma on daily life, 5 point likert scale responses
PROMIS Pediatric Short Form v2.0 - Anxiety | 7 day recall period, taken at the end of each of the four study weeks.
  Short form questionnaire assessing anxiety, 5 point likert scale responses
PROMIS Pediatric Short Form v2.0 - Depressive Symptoms | 7 day recall period, taken at the end of each of the four study weeks.
  Short form questionnaire assessing depressive symptoms, 5 point likert scale responses
PROMIS Pediatric Short Form v2.0 - Fatigue | 7 day recall period, taken at the end of each of the four study weeks.
  Short form questionnaire assessing fatigue, 5 point likert scale responses
PROMIS Pediatric Short Form v2.0 - Mobility | 7 day recall period, taken at the end of each of the four study weeks.
  Short form questionnaire assessing mobility, 5 point likert scale responses
PROMIS Pediatric Short Form v2.0 - Peer Relationships | 7 day recall period, taken at the end of each of the four study weeks.
  Short form questionnaire assessing peer relationships, 5 point likert scale responses

CONTACTS AND LOCATIONS:
Overall Officials: Bryce Reeve, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Univerity of North Carolina at Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
After data collection is complete, PRO data from this project will be shared with the PEPR consortium as required by the funding mechanism for this project. All data will be deidentified and shared by the consortium through the Harvard Dataverse.
Time Frame: 18 months after data collection is complete. No end date.
Access Criteria: Anyone can access the data via the Harvard Dataverse for any type of analyses.

REFERENCES:
- [Derived] Hernandez ML, Lucas N, Mann C, Lin L, Burbank AJ, Brown J, Sims M, Ivins S, Cunningham A, Maciag MC, Akar-Ghibril N, Bennett AV, Phipatanakul W, Reeve BB. Association of step count with PROMIS pediatric health-related quality of life measures in children and adolescents with persistent asthma. J Allergy Clin Immunol Pract. 2021 Jun;9(6):2492-2494. doi: 10.1016/j.jaip.2021.01.046. Epub 2021 Feb 16. No abstract available. PMID 33601050